CLINICAL TRIAL: NCT04167410
Title: Effects of Perioperative Glycemic Management Protocol on Glycemic Outcomes of Type 2 Diabetic Patients Undergoing Major Abdominal Surgery: a Non-Randomized Controlled Study
Brief Title: Effect of Perioperative Glycemia Protocol on Glycemic Outcomes in Diabetic Patients Undergoing Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Pervin Gökay, Doctor of Philosophy, Department of Nursing, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: SBUniversitesi_nursing
Record Dates: First submitted 2019-09-15; First posted 2019-11-18 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Hyperglycemia; Perioperative Complication
Keywords: Perioperative glycaemic management; Nursing; Glycaemic protocol; Glycaemic management; Stress hyperglycaemia; Surgery and diabetes
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): We did not perform any intervention on the patients in the control group. These patients received routine glycaemia control and healthcare provided to diabetic patients undergoing surgical intervention in the department of general surgery.After receiving written informed consent, the first part of the data collection form on the socio-demographic and disease characteristics of the patients were completed face-to-face. The BG levels of the patients and the medications and insulin used for glycaemic control were recorded one night before surgery. The anxiety levels of the patients were evaluated on the morning of surgery using State-Trait Anxiety Inventory . The second part of the data collection form , which included information on glycaemic management, glycaemia levels and the medications and insulin used on the morning of surgery and during surgery, intensive care stay and the clinical period, was filled in by the nurse on the monitoring and anaesthesia forms.
- intervention group (Experimental): Following the introduction of the glycaemic management protocol to the clinic, data on the patients in the intervention group was collected prospectively between June 2018 and December 2018. management was conducted by nurses in line with the protocol. Data on glycaemic management of the intervention group was similar to the control group.the glycaemic management of patients during the perioperative period was conducted by general surgery nurses according to the protoco
  Interventions: Other: glycaemic management protocol implemented to clinic

INTERVENTIONS:
Other: glycaemic management protocol implemented to clinic — Following the introduction of the glycaemic management protocol to the clinic, data on the patients in the intervention group was collected prospectively between June 2018 and December 2018. Data of the patients in the intervention group was collected after the patient applied to the hospital for surgery or just after the decision on surgery was taken. Patients in the intervention group whose HbA1C values exceeded 7% were referred to endocrinology specialists prior to surgery. Glycaemic management of these patients was evaluated at the department of endocrinology and medications or doses of insulin and oral antidiabetics were changed when necessary. Glycaemic management was conducted by nurses in line with the protocolConsequently, the glycaemic management of patients during the perioperative period was conducted by general surgery nurses according to the protocol.
  Arms: intervention group

SUMMARY:
This study evaluated to the effects of a glycaemic control protocol directed by nurses during the perioperative period on glycaemic outcomes in diabetic patients undergoing major abdominal surgery. The study was conducted at the department of general surgery of a research and training hospital.The study included 47 patients who underwent elective major abdominal surgery between September 2017 and December 2018. The number of patients in the intervention and the control groups was 22 and 25, respectively. The glycemia control protocol will be used in the glycemia management of intervention group,routine glycemia management will be used in the control group.

DETAILED DESCRIPTION:
The prevalence of diabetes among the surgical patient population is 10-15%, and surgical operations are administered to diabetic patients more frequently compared to non-diabetic patients. Diabetes or hyperglycaemia in surgical patients increases mortality and morbidity rates during the perioperative period by 50% compared to non-diabetic patients. Maintaining patient blood glucose (BG) levels of within the target range during the surgical period is crucial to prevent postoperative complications. The target BG level has been modified in line with recent scientific findings; institutions (such as the American Diabetes Association), have prepared new guidelines for the management of glycaemia in critically ill and surgical patients. Insulin infusion is the most effective method to control glycaemia in patients with critical disease or in patients about to undergo major surgery. Therefore, current guidelines recommend the use of reliable and practical glycaemia control protocols during insulin infusion. These protocols should be learnt by all members of the team that provide healthcare. Existing studies suggest that glycaemic management protocols are effective methods to achieve the target BG range and decrease the prevalence of hyperglycaemia and hypoglycaemia in critically ill and major surgery patients in a reliable and effective way.

ELIGIBILITY:
Inclusion Criteria;

* Patients were diagnosed with type 2 diabetes
* Patients planned to undergo elective major abdominal surgery

Exclusion Criteria;

* Patients who had diabetes other than type 2 diabetes
* Patient who had a preoperative glycated haemoglobin A1C (HbA1C) value of 8.5% or greater
* Patient planned to undergo surgery related to the pancreas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Rates of hyperglycaemia development | Each participant was followed between 7-10 days postoperatively. Data of the control group was collected within 8 months prospectively. Data of the intervention group was collected within 7 months prospectively.
  Capillary BG > 180 mg/dl refers to hyperglycemia.
Insulin consumption rate | Each participant was followed between 7-10 days postoperatively. Data of the control group was collected within 8 months prospectively. Data of the intervention group was collected within 7 months prospectively.
  Insulin consumption of each participant was calculatedIn in the postoperative period.
Rates of hypoglycaemia development | Each participant was followed between 7-10 days postoperatively. Data of the control group was collected within 8 months prospectively. Data of the intervention group was collected within 7 months prospectively.
  Capillary blood glucose (BG) < 70 mg/dl refers to hypoglycemia.

CONTACTS AND LOCATIONS:
Overall Officials: Pervin Kurtoglu, PhD, Principal Investigator — GulhaneResearch and Training Hospital
Locations (1):
- Gulhane Research and Training Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De identifield individual participant data for all primary and secondary outcomes measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: data will be available within 2 years of study completion
Access Criteria: the data of study will be requested from the principle researcher by mail

REFERENCES:
- [Background] Compton F, Ahlborn R, Weidehoff T. Nurse-Directed Blood Glucose Management in a Medical Intensive Care Unit. Crit Care Nurse. 2017 Jun;37(3):30-40. doi: 10.4037/ccn2017922. PMID 28572099
- [Background] Duggan EW, Carlson K, Umpierrez GE. Perioperative Hyperglycemia Management: An Update. Anesthesiology. 2017 Mar;126(3):547-560. doi: 10.1097/ALN.0000000000001515. PMID 28121636